#### NCT02873221

Study ID: UBR-MD-04

**Title:** A Multicenter, Randomized, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine With or Without Aura

Statistical Analysis Plan Amd 2 Date: 04-Sept-2018

#### 1. Title Page

#### STATISTICAL ANALYSIS PLAN

# A MULTICENTER, RANDOMIZED, OPEN-LABEL EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND TOLERABILITY OF ORAL UBROGEPANT IN THE ACUTE TREATMENT OF MIGRAINE WITH OR WITHOUT AURA

Amendment 2: 2018-09-04

Protocol Number: UBR-MD-04 Amendment 2

Development Phase:

Product Name: Ubrogepant

Study Statistician:

Sponsor: Allergan Pharmaceuticals

2525 Dupont Drive

Irvine, California USA 92612

+1-714-246-4500 +1-800-347-4500

This document is the property of Allergan. and may not—in full or part—be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan.

# 2. Table of Contents

| 1. | Title | Page | | 1 |
|---|---|---|---|---|
| 2. | Tabl | e of Cor | ntents | 2 |
| | 2.1 | List of | f Tables | 3 |
| | 2.2 | List of | f Figures | 5 |
| 3. | List | of Abbro | eviations and Definition of Terms | 6 |
| 4. | Intro | duction | | 8 |
| | 4.1 | Study | Design Summary | 8 |
| | 4.2 | | Objectives and Endpoints | |
| 5. | Stati | stical M | ethodology and Study Endpoints | 13 |
| | 5.1 | | ical Methods Planned in the Protocol and Determination of Sample Size | |
| | | 5.1.1 | Statistical and Analytical Plans | 13 |
| | | | 5.1.1.1 Common Conventions | |
| | | | 5.1.1.2 Demographics | 18 |
| | | | 5.1.1.4 Safety Analyses | 2.0 |
| | | | 5.1.1.4 Safety Analyses | |
| | | | 5.1.1.6 Interim Analyses | |
| | 5.2 | Chang | ges in the Conduct of the Study or Planned Analyses | 35 |
| | | 5.2.1 | Changes in the Conduct of the Study | 35 |
| | | 5.2.2 | Changes to Analyses Prior to Database Lock | |
| 6. | Data | Handlir | ng and Analysis Conventions | 36 |
| | 6.1 | Study | Treatment Conventions | 36 |
| | | 6.1.1 | Analysis Days | 36 |
| | | 6.1.2 | Missing/Incomplete Treatment End Date | 36 |
| | 6.2 | Analy | sis Visit Windows | 36 |
| | | 6.2.2 | Safety | 37 |

| | | 625 | 6.3.4.2 | AE Group of Interest | |
|---|---|---|---|---|---|
| | | 6.3.5 | | Laboratory Assessments | |
| | | | 6.3.5.1 | Potentially Clinically Significant Criteria | |
| | | | 6.3.5.2<br>6.3.5.3 | Hepatic Laboratory Abnormalities Continuous Descriptives and Shift Table Parameters | |
| | | | 6.3.5.4 | Character Values | |
| | | 6.3.6 | | gns | |
| | | 0.5.0 | 6.3.6.1 | Potentially Clinically Significant Criteria | |
| | | | 6.3.6.2 | Continuous Descriptives and Shift Table Parameters | |
| | | 6.3.7 | Electroc | ardiograms | |
| | | | 6.3.7.1 | QTc Derivation | 45 |
| | | | 6.3.7.2 | Potentially Clinically Significant Criteria | 45 |
| | | | 6.3.7.3 | Continuous Descriptives and Shift Table Parameters | |
| | 6.4 | Impute | ed Value I | Listing Conventions | 46 |
| 7. | Ame | ndment( | (s) | | 46 |
| 8. | Appe | pendices | | | |
| ٠. | 8.1 | | | ferred Terms for AE Categories of Clinical Interest Created by S | |
| 2. | 1 | ī | ist of Ta | ahles | |
| | | | | | _ |
| Tal | ble 3-1 | A | bbreviatio | ons and Definitions of Terms | 6 |
| Tal | ble 4-1 | S | tudy Objec | ctives and Corresponding Endpoints | 9 |
| Tal | ble 5-1 | A | nalysis Po | opulations | 13 |
| Tal | ble 5-2 | S | tatistical N | Methodology | 14 |
| Tal | ble 5-3 | N | lissing Da | ta Handling by Endpoint Type | 15 |
| Tal | ble 5-4 | A | nalysis Po | opulation Summaries | 18 |
| Tal | ble 5-5 | P | articipant i | Disposition Summaries | 18 |
| | ble 5-6 | | • | on of Renal Function Based on Estimated GFR (eGFR) | |
| | ble 5-7 | | | eviation Summary | |
| | | | | • | |
| Ta | ble 5-8 | D | emograph | ic Summaries | 20 |

| Table 5-9 | Baseline Characteristics Summaries | 20 |
|---|---|---|
| Table 5-10 | Medical History Summary | 21 |
| Table 5-11 | Migraine History Summary | 21 |
| Table 5-12 | Medication Summaries | 22 |
| Table 5-16 | Safety Endpoint Baseline Definitions | 26 |
| Table 5-17 | Treatment Exposure Summaries | 27 |
| Table 5-18 | Treatment Compliance Summaries | 28 |
| Table 5-19 | AE Terms | 28 |
| Table 5-20 | AE Summaries | 29 |
| Table 5-21 | Clinical Laboratory Summaries | 31 |
| Table 5-22 | Potential Hy's Law Summaries | 32 |
| Table 5-23 | Vital Signs Summaries | 32 |
| Table 5-24 | ECG Summaries | 33 |
| Table 5-25 | Cardiovascular Risk Summaries | 34 |
| Table 5-26 | Suicidality Summaries | 34 |
| Table 6-1 | Analysis Day Definitions | 36 |
| Table 6-4 | Safety Analysis Visit Definitions for 3-Month Time Interval | 37 |
| Table 6-5 | Safety Analysis Visit Definitions for 1-Month Time Interval | 37 |
| Table 6-6 | Safety Analysis Visit Definitions | 37 |
| Table 6-10 | Construction Methods for AE Categories of Clinical Interest | 40 |

| 2.2 | List of Figures |
|---|---|
| Table 8-2 | List of Preferred Terms for Hepatic Disorder Broad SMQ |
| Table 8-1 | List of Preferred Terms for AE Categories of Clinical Interest Created by Narrow SMQs. |
| Table 6-19 | ECG Descriptive and Shift Table Parameters46 |
| Table 6-18 | ECG PCS Criteria 46 |
| Table 6-17 | QTc Derivation |
| Table 6-16 | Vital Sign Descriptive and Shift Table Parameters |
| Table 6-15 | Vital Sign PCS Criteria |
| Table 6-14 | Clinical Descriptive and Shift Table Parameters |
| Table 6-13 | Criteria for Hepatic Laboratory Abnormalities |
| Table 6-12 | Clinical Laboratory PCS Criteria |
| Table 6-11 | Preferred Terms for Abuse-Related Category and Triptan-Associated Category41 |

# 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Tubic o T | Appreviations and Definitions of Terms |
|---|---|
| Abbreviation/Term | Definition |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | body mass index |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CFB | change from baseline |
| CHD | coronary heart disease |
| CSR | clinical study report |
| CV | cardiovascular |
| eCRF | electronic case report form |
| ECG | electrocardiogram, electrocardiographic |
| FDS | Functional Disability Scale |
| HEOR | Health Economics and Outcomes Research |
| INR | international normalized ratio |
| IWRS | interactive web response system |
| kg | kilogram(s) |
| LOCF | last observation carried forward |
| m | meter(s) |
| MedDRA | Medication Dictionary for Regulatory Activities |
| mg | milligrams |
| mITT | modified intent-to-treat |
| MQoLQ | migraine quality of life questionnaire |
| PCS | potentially clinically significant |
| PF | pain free |
| PK | pharmacokinetic |
| PR | pain relief |
| PT | preferred term |
| QTc | QT interval corrected for heart rate |
| QTcB | QT interval corrected for heart rate using the Bazett formula $(QTcB = QT/(RR)^{\frac{1}{2}})$ |
| QTcF | QT interval corrected for heart rate using the Fridericia formula $(QTcF = QT/(RR)^{\frac{1}{3}})$ |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Statistical Analysis Software |
| SD | standard deviation |
| SE | standard error |
| 1- | |

| Abbreviation/Term | Definition |
|---|---|
| SI | Le Système International d'Unités (International System of Units) |
| SOC | system organ class |
| SPF | sustained pain freedom |
| TBL | total bilirubin |
| TEAE | treatment-emergent adverse event |
| ULN | upper limit of normal |
| US | United States of America |
| WHO | World Health Organization |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the efficacy and safety data outlined and/or specified in the protocol amendment #2 dated 06 Dec 2017 of Study UBR-MD-04. Specifications of tables, figures, and data listings are contained in a separate document. The SAP for health economics and outcomes research (HEOR) data will be prepared separately.

This document is organized into 3 main sections:

- 1. Study overview
- 2. Statistical Methodology and Study Endpoints
- 3. Data Handling and Analysis Conventions

#### 4.1 Study Design Summary

*Structure:* Multicenter, randomized, open-label, 52-week extension study; randomization to the ubrogepant arms (50 and 100 mg) will be blinded.

Duration: 52 weeks

Study Treatment Groups: usual care, ubrogepant 50 mg, or ubrogepant 100 mg

Controls: Not applicable

Dosage/Dose Regimen: Patients randomized to either of the ubrogepant arms will treat up to 8 migraine attacks (of any pain severity) every 4 weeks at home for a total 1 year. Patients have the option to take a second dose of ubrogepant if the patient has either a nonresponding migraine or a migraine recurrence. The second dose of ubrogepant will be identical to the first dose.

Patients randomized to the usual-care arm will be instructed to treat their migraine with medications that they routinely use to relieve a migraine attack.

Randomization/Patients will be randomized (1:1:1) to 1 of the following 3 treatment groups: usual care, ubrogepant 50 mg, or ubrogepant 100 mg. The study is open-label; however, randomization to the ubrogepant arms (50 and 100 mg) will be blinded.

*Number of Participants:* Approximately 1200 patients will be randomized (400 patients per arm) from approximately 200 centers in the United States.

#### 4.2 Study Objectives and Endpoints

Each study objective is presented with corresponding endpoint(s) below:

Table 4-1 Study Objectives and Corresponding Endpoints

# **Objectives Endpoints Primary** • [PO1] To evaluate the safety and tolerability of intermittent treatment with ubrogepant for the acute treatment of migraine over 1 year



# 4.3 Schedule of Activities



#### 5. Statistical Methodology and Study Endpoints

# 5.1 Statistical Methods Planned in the Protocol and Determination of Sample Size

This statistical analysis plan (SAP) will be approved prior to database lock. The SAP expands the statistical section of the protocol and contains a detailed description of methods to analyze data collected in the study. The text portion of the SAP will be included in the clinical study report (CSR) report as Appendix 16.1.9.

#### 5.1.1 Statistical and Analytical Plans

Statistical analyses will be conducted using

#### **5.1.1.1** Common Conventions

#### 5.1.1.1.1 Analysis Populations

The analysis populations will consist of participants as defined below:

Table 5-1 Analysis Populations

| Population | Definition | Study Treatment |
|---|---|---|
| Screened | All screened participants who signed informed consent | _ |
| Intent-to-Treat (ITT) | All randomized participants. | Randomized assignment |
| Modified Intent-to- | All randomized patients who received at least 1 dose of IP | Randomized assignment |
| Treat (mITT) | (ubrogepant) and had at least 1 posttreatment efficacy assessment | |
| | in this study. The mITT population is only defined for the | |
| | ubrogepant arms, as no posttreatment efficacy measurements will | |
| | be collected from patients in the usual-care arm. | |
| Safety | The Safety population is defined separately below for the | Actual received |
| | ubrogepant arms and the usual-care arm. | |
| | Ubrogepant arms: All randomized patients who received $\geq 1$ dose of treatment. | |
| | Usual care arm: All randomized patients in the usual-care arm. | |
| | The purpose of the usual care arm is to contextualize any safety findings that may occur in the ubrogepant treated patients over the course of 12 months. As such, data from all patients randomized to the usual care arm, regardless of whether the patient used medication to treat migraine, will be included in the safety analyses. | |

### **5.1.1.1.2** Study Treatments

The following treatment groups are defined for this study:

- Usual Care
- Ubrogepant 50 mg
- Ubrogepant 100 mg

## 5.1.1.1.3 Statistical Methodology

The methodologies defined below apply as specified to individual endpoints defined in this SAP. All statistical tests will be 2-sided hypothesis tests performed at the 5% level of significance for main effects. All confidence intervals will be 2-sided 95% confidence intervals, unless stated otherwise.

Table 5-2 Statistical Methodology

| Methodology | | Description |
|---|---|---|
| M1 | Categorical | Number of participants in individual categories |
| | counts | o Participants with ≥ 1 qualifying event counted once per individual category |
| M2 | Categorical descriptives | <ul> <li>Number and percentage of participants in individual categories <ul> <li>○ Participants with ≥ 1 qualifying event counted once per individual category</li> </ul> </li> <li>N1 if proportion denominator ≠ number of participants in the population (standard percentage denominator)</li> <li>○ N1 = participants with non-missing baseline value</li> </ul> |
| M3 | PCS<br>descriptives | Number and percentage of participants meeting potentially clinically significant |
| M4 | Shift<br>analysis | <ul> <li>Number and percentage of participants in individual baseline and postbaseline categories</li> <li>Percentage denominator = number of participants in individual baseline categories</li> <li>N1 = participants with non-missing values at both baseline and the specified postbaseline analysis visit</li> </ul> |
| M5 | Continuous descriptives | <ul> <li>N1, mean, standard deviation (SD), median, minimum, maximum</li> <li>N1 = participants with non-missing value</li> </ul> |
| M6 | CFB descriptives | <ul> <li>Continuous descriptives for baseline, postbaseline, and change from baseline (CFB) values</li> <li>N1 = participants with non-missing values at both baseline and the specified postbaseline analysis visit</li> </ul> |
| M7 | Responder | <ul> <li>Categorical descriptives using proportions for responders and nonresponders <ul> <li>Nonresponders include:</li> <li>Participants who do not meet responder criteria</li> </ul> </li> <li>N1 = all participants unless otherwise specified</li> </ul> |
| M8 | Logistic<br>regression<br>model | Measures the relationship between the binomial dependent variable (number of events among number of treated attacks) and independent variables: |

| Methodology | Description |
|---|---|
| | <ul> <li>Odds ratio for comparing the percentage of treated attacks with PF at 2 hours for a</li> </ul> |
| | given 3-month interval with that for the first 3-month interval and its 95% |
| | confidence interval will be derived from the mixed logistic regression model for |
| | each of the 2 ubrogepant treatment groups. |
| | <ul> <li>Calculate two-sided p-values</li> </ul> |

CFB = change from baseline.

Raw and derived data listings will be provided, and will be fully defined in the table, figure, and data listing specification document.

#### **5.1.1.1.4 Missing Data**

General missing data handling conventions are specified for methodologies in Section 5.1.1.1.3 and summarized as follows:

Table 5-3 Missing Data Handling by Endpoint Type

| Parameter type | Timing | Missing Data Handling |
|---|---|---|
| Responder | Treatment Period | • If missing headache severity, migraine-associated symptoms, |
| | | use Observed Cases (OC) |

A conservative approach will used to resolve the incompatibility between the answers to the headache recurrence questions at the 24- and 48-hour time points for each treated attack by setting the answer to the recurrence question at the 48-hour time point the same as the answer to the recurrence question at the 24-hour time point recurrence question indicates headache recurrence between 2 and 24 hours but the 48-hour time point recurrence question indicates either no or a less severe headache recurrence between 2 and 48 hours for the same treated attack.







### 5.1.1.2 Demographics

#### 5.1.1.2.1 Analysis Populations

The distribution of participants within the analysis populations will be summarized as follows:

Table 5-4 Analysis Population Summaries

| Population | Description | Timing | Methodology |
|---|---|---|---|
| Screened Population | Distribution overall and within sites in | | Categorical counts |
| | total | | |
| | Distribution by lead-in study treatment and | | |
| | within extension study in total | | |
| ITT, mITT, and Safety | Distribution overall and within sites in | _ | Categorical counts |
| populations | total and by treatment group | | |
| | Distribution by lead-in study treatment and | | |
| | by extension study treatment | | |

#### **5.1.1.2.2** Participant Disposition

Participant disposition encompasses the distribution of participants who enter, complete, and discontinue each specified analysis period, along with eCRF-reported discontinuation reasons from each respective analysis period. Participant disposition will also be presented for the relevant subgroups including sex, age group, race, CV risk category, and renal function class. The subgroups are defined in the lead-in studies. Participant disposition will be summarized as follows:

Table 5-5 Participant Disposition Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Screening disposition <sup>1</sup> | Distribution in the Screened Population in | Screening Period | Categorical |
| | total | | descriptives |
| Treatment disposition | Distribution in the Safety Population and ITT Population in total and by treatment group for all participants and by subgroups: • by sex, • by age group (<40 years vs ≥40 years) • by age subgroup (<65 years vs ≥65 years) • by race (white vs non-white) • by cardiovascular risk category (high risk, moderate risk, and low risk) • by renal function class (normal, | Treatment Period | Categorical descriptives |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | mild renal impairment, moderate | | |
| | renal impairment) | | |
| 4 Week Safety Follow-<br>up disposition <sup>1</sup> | Distribution in the Safety Population and ITT Population in total and by treatment group for all participants and by subgroups: • by sex, • by age group (<40 years vs ≥40 years) • by age subgroup (<65 years vs ≥65 years) • by race (white vs non-white) • by cardiovascular risk category (high risk, moderate risk, and low risk) • by renal function class (normal, mild renal impairment, moderate renal impairment) | Post-treatment Period | Categorical descriptives |

Participant disposition will be listed and participants who prematurely discontinued will be listed.

CV risk subgroup will be derived as a categorical variable with three categories based on NCEP ATP III: Category 1 (High Risk): > 20% 10-year CV risk, Category 2 (Moderate Risk): 10 - 20% 10-year CV risk, and Category 3 (Low Risk): <10% 10-year CV risk.

Renal function class will be derived as a categorical variable based on baseline eGFR as shown in Table 5-6. Since only a few participants are classified into the categories of severe renal impairment or ESRD, renal function class for subgroup analyses will focus on the following categories: Normal, Mild renal impairment, Moderate renal impairment. A listing of all AEs for participants with severe renal impairment or ESRD will be provided including treatment group, participant ID, study center, and baseline eGFR.

Table 5-6 Classification of Renal Function Based on Estimated GFR (eGFR)

| Stage | Renal Function Class | eGFR <sup>a</sup> (mL/min/1.73m <sup>2</sup> ) |
|---|---|---|
| 1 | Normal | ≥ 90 |
| 2 | Mild renal impairment | 60-89 |
| 3 | Moderate renal impairment | 30-59 |
| 4 | Severe renal impairment | 15-29 |
| 5 | End Stage Renal Disease (ESRD) | <15 not on dialysis |

<sup>&</sup>lt;sup>a</sup> eGFR: estimate of GFR based on a Modification of Diet in Renal Disease (MDRD) equation.

#### 5.1.1.2.3 Protocol Deviations

Protocol deviations will be defined in Protocol Deviation Requirement Specification, including importance classification. Protocol deviations will be summarized as follows:

Table 5-7 Protocol Deviation Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Major protocol | Distribution in the ITT Population in total | _ | Categorical |
| deviations <sup>1</sup> | and by treatment group | | descriptives |

<sup>&</sup>lt;sup>1</sup> Protocol deviations will be listed.

#### 5.1.1.2.4 Demographics

Demographics will be summarized in total and by treatment group for the ITT, Safety, and mITT populations, as follows:

Table 5-8 Demographic Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Age <sup>1</sup> | Age (years) relative to informed consent | Informed consent in | Continuous |
| | date | the lead-in study | descriptives |
| Age group | Age group 1: | Informed consent in | Categorical |
| | • <20 | the lead-in study | descriptives |
| | • 20 to 29 | | |
| | • 30 to 39 | | |
| | • 40 to 49 | | |
| | • 50 to 59 | | |
| | • 60 to 69 | | |
| | • ≥ 70 | | |
| | Age group 2: | | |
| | • <40 | | |
| | • ≥40 | | |
| | Age group 3: | | |
| | • <65 | | |
| | • ≥65 | | |
| Sex, race, and ethnicity <sup>1</sup> | eCRF categories | Screening Period in | Categorical |
| | Race group | the lead-in study | descriptives |
| | o White | | |
| | o Non-white | | |

<sup>&</sup>lt;sup>1</sup> Participant demographics will be listed.

#### **5.1.1.2.5** Baseline Characteristics

Baseline characteristics will be summarized in total and by treatment group for the ITT, Safety, and mITT populations as follows:

Table 5-9 Baseline Characteristics Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Baseline characteristics <sup>1</sup> | • Height (m) | Latest assessment in | Continuous |
| | • Weight (kg) | Screening Period in | descriptives |
| | Body mass index (BMI) | the lead-in study | |
| | • Weight (kg) / height (m) <sup>2</sup> | | |
| Cardiovascular risk <sup>2</sup> | Cardiovascular risk factor subgroup | Randomization date | Categorical |
| | • low risk | in the lead-in study | descriptives |
| | <ul> <li>moderate risk</li> </ul> | | |
| | <ul> <li>high risk</li> </ul> | | |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Renal function class <sup>2</sup> | Renal function class subgroup | Randomization date | Categorical |
| | <ul> <li>Normal</li> </ul> | in the lead-in study | descriptives |
| | <ul> <li>Mild renal impairment</li> </ul> | | |
| | Moderate renal impairment | | |
| Randomization strata <sup>3</sup> | Previous response to triptans | Randomization date | Categorical |
| | <ul> <li>Triptan Responder</li> </ul> | in the lead-in study | descriptives |
| | <ul> <li>Triptan Insufficient Responder</li> </ul> | | |
| | Triptan Naïve | | |
| | Triptan Insufficient Responder will be | | |
| | further classified into subcategories | | |
| | <ul> <li>Insufficient Efficacy</li> </ul> | | |
| | <ul> <li>Insufficient Tolerability</li> </ul> | | |
| | <ul> <li>Contraindications/Warnings or</li> </ul> | | |
| | Precautions | | |
| | Current use of prophylactic concomitant | | |
| | medication for migraine (Yes, No) | | |

<sup>&</sup>lt;sup>1</sup> Participant baseline characteristics will be listed.

#### 5.1.1.2.6 Medical History

Medical history, encompassing abnormalities and surgeries reported as occurring before the Screening Visit in the lead-in study, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 20.1 or newer. Unique participants who report medical history events will be summarized by MedDRA system organ class (SOC) and preferred term (PT) in total and by treatment group for the Safety Population as follows:

Table 5-10 Medical History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Medical history <sup>1</sup> | Abnormalities and surgeries occurring | Screening Period in | Categorical |
| | before the Screening Visit by treatment | the lead-in study | descriptives |
| | group | | |

SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group.

# 5.1.1.2.7 Migraine History

Migraine history (based on the lead-in study), including diagnosis, duration of disorder, previous use of prophylaxis treatment, average frequency of moderate to severe migraines per month in past 3 months, and acute treatments will be reported in total and by treatment group for the Safety Population as follows:

Table 5-11 Migraine History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Migraine Diagnosis <sup>1</sup> | With Aura | Screening Period | Categorical |
| | Without Aura | in the lead-in | descriptives |
| | • Both | study | |
| Previous Prophylaxis | Yes or No | Screening Period | Categorical |
| Migraine Treatment <sup>1</sup> | | in the lead-in | descriptives |
| | | study | |
| Acute Migraine | Categorize as Yes or No, and | Screening Period | Categorical |
| Treatment <sup>1</sup> | subcategorize the Yes by: | in the lead-in | descriptives |

<sup>&</sup>lt;sup>2</sup> Summary for Safety population only.

<sup>&</sup>lt;sup>3</sup> Participant randomization scheme and codes will be listed.

<sup>&</sup>lt;sup>1</sup> Participant medical history will be listed.

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | Triptan | study | |
| | <ul> <li>Ergot or Ergot Combinations</li> </ul> | | |
| | NSAID | | |
| | Opiate or Opiate Combination | | |
| | Antiemetic Agent | | |
| | Barbiturates | | |
| | • Other | | |
| Migraine Disorder | In the Table summarize in Years, in the | Screening Period | Continuous |
| Duration <sup>1</sup> | Listing show original data in Years and | in the lead-in | descriptives |
| | Months | study | |
| Average Frequency of | N/A | Screening Period | Continuous |
| Moderate to Severe | | in the lead-in | descriptives |
| Migraines per Month in | | study | |
| Last 3 Months | | | |

<sup>&</sup>lt;sup>1</sup>Participant migraine history will be listed.

#### **5.1.1.2.8** Prior and Concomitant Medications

Medications will be coded using the World Health Organization (WHO) Drug Dictionary, version March 2016 or newer. Unique participants who reported medications will be summarized by Anatomical Therapeutic Chemical (ATC) 4 class and PT in total and by treatment group for the Safety Population as follows:

**Table 5-12 Medication Summaries** 

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Prior medications <sup>1</sup> | Medications taken $\geq 1$ time before the | Screening Period in | Categorical |
| | study treatment start date of the lead-in | the lead-in study | descriptives |
| | study, regardless of medication end date | | |
| Concomitant | Medications taken $\geq 1$ time on or after the | Treatment Period | Categorical |
| medications <sup>1</sup> | randomization date, regardless of | | descriptives |
| | medication start date | | |

ATC4 classes will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group. 

1 Participant prior and concomitant medication will be listed.











#### **5.1.1.4** Safety Analyses

Safety analyses will be based on the Safety Population.

Baseline assessments for applicable safety endpoints are defined as follows:

Table 5-16 Safety Endpoint Baseline Definitions

| Parameter | Description | Timing |
|---|---|---|
| Clinical laboratory evaluations | eCRF- or (standardized) vendor-provided | Latest non-missing |
| <ul> <li>Vital signs</li> </ul> | assessments | assessment before the first |
| • Electrocardiograms (ECGs) | | dose of treatment in the |
| | | lead-in study |

### 5.1.1.4.1 Study Treatment Exposure and Compliance

Study treatment exposure will be listed for the Safety Population.

The listing of treatment exposure will indicate whether the participant took the optional second dose in addition to the first dose for each attack.

For safety analyses only, the number of treated migraine attacks will be determined based on the date and time (if available from eDiary) doses were taken. Starting with the first dose taken by each participant, doses will be sorted based on the date and time (if available from eDiary) each dose was taken. Subsequent doses that are separated by at least 2 calendar days or 48 hours will be considered the initial treatment for a separate and distinct migraine attack. Doses taken within the 2-calendar day/48-hour window of the initial dose will be considered as additional doses treating the same attack. As such, the treatment label (initial dose or optional second dose) will be ignored. The extent of exposure to study treatment will be summarized as follows:

Table 5-17 Treatment Exposure Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Number of participants | For all participants: | Treatment period | Categorical |
| with study participation | • total number (%) of participants | | descriptives |
| by 3-month interval | who completed 3 months | | |
| | • total number (%) of participants | | |
| | who completed 6 months | | |
| | • total number (%) of participants | | |
| | who completed 9 months | | |
| | <ul> <li>total number (%) of participants</li> </ul> | | |
| | who completed 12 months | | |
| | Subgroup analyses: | | |
| | • by Sex | | |
| | <ul> <li>by Age Group: &lt;40 vs ≥40</li> </ul> | | |
| | 1 2 2 | | |
| | by Race White vs All other races | | |
| | by CV risk category | | |
| 27 1 2 | by renal function class | | |
| Number of participants | • total number (%) of participants | Treatment period | Categorical |
| with study participation | who completed 3 months | | descriptives |
| by 3-month interval | • total number (%) of participants | | |
| among those who | who completed 6 months | | |
| treated at least 2 | • total number (%) of participants | | |
| migraine attacks per | who completed 9 months | | |
| month on average | • total number (%) of participants | | |
| during the completed | who completed 12 months | | |
| interval | | T | <u> </u> |
| Number of migraine | total number of migraine attacks | Treatment period | Continuous |
| attacks treated over the | treated with only one dose | | descriptives |
| entire duration of the study <sup>1</sup> | • total number of migraine attacks | | |
| study | treated with two or more doses | | |
| N. 1. 0 1 | total number of doses taken | T | <u> </u> |
| Number of attacks | • >= 8 | Treatment period | Categorical |
| treated with study | $\bullet$ >= 6 and < 8 | | descriptives |
| treatment per month <sup>1</sup> | $\bullet$ >= 4 and < 6 | | |
| | $\bullet$ >= 2 and < 4 | | |
| | • <2 | | |
| Average number of | For all participants: | Treatment period | Categorical |
| attacks treated with | • >= 8 | | descriptives |
| study treatment per | $\bullet$ >= 6 and < 8 | | |
| month <sup>1</sup> | $\bullet$ >= 4 and < 6 | | |
| | $\bullet$ >= 2 and < 4 | | |
| | • <2 | | |
| | Subgroup analyses: | | |
| | • by Sex | | |
| | • by Age Group: <40 vs ≥40 | | |
| | <ul> <li>by Age Group: &lt;65 vs ≥65</li> </ul> | | |
| | <ul> <li>by Race White vs All other races</li> </ul> | | |
| | <ul> <li>by CV risk category</li> </ul> | | |
| | <ul><li>by renal function class</li></ul> | | |
| Maximum number of | • >= 8 | Treatment period | Categorical |
| attacks treated with | • >= 6 and < 8 | Troumfont period | descriptives |
| study treatment per | | | acceripe ( es |
| stady incuminant per | $\bullet$ >= 4 and < 6 | | |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| month, defined as maximum of monthly total number attacks treated with study treatment among months 1-12 for each participant <sup>1</sup> | <ul><li>&gt;= 2 and &lt; 4</li><li>&lt; 2</li></ul> | | |
| Number of months with<br>the number of attacks<br>treated with study<br>treatment in each<br>category <sup>1</sup> | For each category: • >= 8 • >= 6 and < 8 • >= 4 and < 6 • >= 2 and < 4 • < 2 | Treatment period | Categorical<br>descriptives |
| Average number of study treatment taken per month <sup>1</sup> | <ul> <li>&gt;= 16</li> <li>&gt;= 14 and &lt; 16</li> <li>&gt;= 12 and &lt; 14</li> <li>&gt;= 10 and &lt; 12</li> <li>&gt;= 8 and &lt; 10</li> <li>&gt;= 6 and &lt; 8</li> <li>&gt;= 4 and &lt; 6</li> <li>&gt;= 2 and &lt; 4</li> <li>&lt; 2</li> </ul> | Treatment period | Categorical descriptives |

Analysis visits defined in Section 6.2.2.

Treatment compliance for this study will be summarized as follows:

Table 5-18 Treatment Compliance Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Overdosing <sup>1</sup> | Participants who took more than 2 doses | | Listing |
| | within 48 hours or 2 calendar days (if time | | |
| | information is not available) | | |
| | · | | |

<sup>&</sup>lt;sup>1</sup> Participants in the ubrogepant treatment arms only.

#### 5.1.1.4.2 Adverse Events

The following adverse event (AE) terms are defined:

Table 5-19 AE Terms

| Term | Description |
|---|---|
| Treatment- | An event that initially occurs or increases in intensity on or after the initial dose of treatment of |
| emergent | the lead-in study. An event that occurs after Visit 16 for participants with Visit 16, or more than |
| | 30 days after the last visit or last treatment, whichever is later, for participants without Visit 16 |
| | will not be considered as treatment-emergent. |

<sup>&</sup>lt;sup>1</sup> Participants in the ubrogepant treatment arms only. No imputation for the last incomplete month.

| Term | Description |
|---|---|
| On-therapy | An event where: |
| | • Treatment start date of the lead-in study ≤ event start date ≤ Visit 16 for participants with Visit 16, or within 30 days after the last visit or last treatment, whichever is later, for participants without Visit 16 |

AEs, encompassing abnormalities and surgeries reported as occurring after the Screening Visit, will be coded using MedDRA version 20.1 or newer. Unique participants reporting AEs in the following AE categories will be summarized by treatment group for the Safety Population as follows:

Table 5-20 AE Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Overall summary | Overall summary only for the following | From randomization date | Categorical |
| | categories: | to Visit 16 for participants | descriptives |
| | Treatment-emergent AEs | with Visit 16, or within 30 | P |
| | (TEAEs) | days after last visit or last | |
| | <ul> <li>Treatment-related TEAEs</li> </ul> | treatment, whichever is | |
| | <ul> <li>On-therapy serious adverse events</li> </ul> | later, for participants | |
| | (SAEs) | without Visit 16 | |
| | • Deaths | | |
| | <ul> <li>AEs leading to discontinuation</li> </ul> | | |
| | Subgroup analyses by Cardiovascular Risk | | |
| | Category and by renal function class | | |
| TEAEs | Summary by | From randomization date | Categorical |
| TEAES | SOC and PT for all participants | to Visit 16 for participants | descriptives |
| | and by subgroup analyses: | with Visit 16, or within 30 | descriptives |
| | o by Sex | days after last visit or last | |
| | o by Age Group <40 vs | treatment, whichever is | |
| | o by Age Gloup <40 vs<br>≥40 | later, for participants | |
| | o by Age Group <65 vs | without Visit 16 | |
| | 0 by Age Gloup <05 vs<br>≥65 | Without Visit 10 | |
| | o by Race White vs All | | |
| | other races | | |
| | o by cardiovascular risk | | |
| | category | | |
| | o by renal function class | | |
| | SOC and PT for concomitant | | |
| | medication classes used by at | | |
| | least 10% of participants in at | | |
| | least one treatment group | | |
| | • SOC, PT, and AE onset time | | |
| | intervals | | |
| | ○ <3 months | | |
| | $\circ$ $\geq$ 3 and $\leq$ 6 months | | |
| | $\circ \ge 6$ and $< 9$ months | | |
| | $\circ \ge 9$ and $\le 12$ months | | |
| | $\circ \ge 12 \text{ months}$ | | |
| | <ul> <li>SOC, PT, and average number of</li> </ul> | | |
| | migraine attacks treated with | | |
| | study treatment per month | | |
| | o ≥2 | | |
| | o ≥4 | | |
| | o ≥6 | | |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | <ul> <li>≥8</li> <li>SOC, PT, and severity</li> <li>SOC, PT, and causal relationship to the study treatment</li> <li>Type (Mild, Moderate, Severe, related, not related)</li> <li>SOC and PT for TEAEs occurring in ≥ 2% of participants in any ubrogepant treated dose group (and greater than placebo)</li> </ul> | | |
| Common TEAEs | Summary by PT • Includes TEAEs occurring in ≥ 2% of participants in any treatment group | From randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16 | Categorical<br>descriptives |
| On-therapy SAEs <sup>1</sup> | Overall summary and by PT | From randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16 | Categorical descriptives |
| On-therapy fatal SAEs | Participants who report On-therapy fatal SAEs will have their fatal SAEs and all AEs listed | From randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16 | Categorical descriptives |
| AEs leading to discontinuation <sup>2</sup> | Overall summary and by PT | From randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16 <sup>2</sup> | Categorical<br>descriptives |
| TEAEs of specific interest <sup>3</sup> | Overall summary and by PT for the following type of TEAEs: • Hepatic Injury TEAEs • Cardiac Arrhythmias TEAEs • Central Nervous System Vascular Disorders TEAEs • Embolic and Thrombotic Events TEAEs • Hypertension TEAEs • Hypertension TEAEs • Ischaemic Heart Disease TEAEs • Suicide/self-injury TEAEs • Triptan-associated TEAEs • Abuse-related TEAEs | From randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16 | Categorical<br>descriptives |

SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose group. If more than 1 AE is coded to the same participant, the participant will be counted only once for that preferred term using the greatest severity

Parameter Description Timing Methodology

If more than 1 AE is coded to the same participant, the participant will be counted only once for that preferred term using the strictest causal relationship to treatment for the summarization by causal relationship

#### **5.1.1.4.3** Clinical Laboratory Assessments

Clinical laboratory assessments will be summarized by treatment group for the Safety Population as follows:

Table 5-21 Clinical Laboratory Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Number and percentage<br>of participants with<br>Potentially Clinically<br>Significant (PCS)<br>values <sup>1</sup> | Summary by laboratory category, parameter, and PCS criteria • Parameters and PCS criteria specified in Section 6.3.5.1 • N1 (percentage denominator) = Participants with non-missing non-PCS baseline and >=1 postbaseline parameter assessment | Randomization to<br>End of Study <sup>3</sup> | PCS descriptives |
| Descriptives <sup>2</sup> | Summary by laboratory category and parameter in SI units and in conventional units and analysis visit • Parameters specified in Section 6.3.5.3 | Randomization to<br>End of Study <sup>3</sup> | CFB descriptives |
| Shift from baseline | Summary by laboratory parameter and category • Low, normal, and high categories provided by central laboratory • Parameters specified in Section 6.3.5.3 | End of Study <sup>3</sup> | Shift analysis |
| Liver function findings <sup>4</sup> | Summary of number and percentage by hepatic laboratory parameter and PCS categories. Definition of PCS categories see Table 6-10 in Section 6.3.4.2. | Randomization to<br>End of Study <sup>3</sup> | Categorical descriptives |
| Adjudication results of ALT or AST elevations <sup>5</sup> | Summary of relationship of ALT or AST elevation to study medication for participants with adjudicated case (i.e., ALT ≥ 3xULN and/or AST ≥ 3xULN) by the following categories: • Probable • Possible • Unlikely • Insufficient data Summary will be provided for the incidence by number of participants and by number of events | Randomization date<br>to End of Study <sup>3</sup> | Categorical descriptives |

ALT = aspartate aminotransferase; AST = aspartate aminotransferase; TBL = total bilirubin; ALP = alkaline phosphatase; INR = international normalized ratio; ULN = upper limit of normal.

<sup>&</sup>lt;sup>1</sup> Participants who report  $\geq$  1 SAE will have their SAE listed.

<sup>&</sup>lt;sup>2</sup> If the discontinued date is from randomization date to Visit 16 for participants with Visit 16, or within 30 days after last visit or last treatment, whichever is later, for participants without Visit 16, then AEs leading to discontinuation will be summarized and listed

<sup>&</sup>lt;sup>3</sup> Participants who reported  $\geq 1$  AEs in the corresponding category will have these AEs listed.

<sup>&</sup>lt;sup>1</sup> Participants who report ≥ 1 postbaseline PCS value will have their laboratory visits with PCS values and all AEs listed.

<sup>&</sup>lt;sup>2</sup>Clinical laboratory results and comments will be listed.

<sup>&</sup>lt;sup>3</sup> Analysis visits defined in Section 6.2.2.

| Endpoint | Description | Timing | Methodology |
|----------|-------------|--------|-------------|

<sup>&</sup>lt;sup>4</sup> Details of all participants with any liver function laboratory findings will be listed. For participants who met  $ALT \ge 3xULN$  or  $AST \ge 3xULN$ , their ALT, AST, TBL, ALP, and INR assessments, and all AEs will be listed for all study visits. In addition, if available, their abnormal liver biochemistries risk factors, liver disease signs and symptoms, liver diagnostic tests, specialist consultation, liver lab tests, and drug screen will also be listed.

Evaluation of drug-induced serious hepatoxicity (eDISH) plot (scatter plot of maximum total bilirubin vs. maximum ALT) will be generated. The ALT, AST, total bilirubin, and ALP values over time will be overlaid on the same plot along with indicators for dosing times for each participant with ALT or AST elevation ( $\geq 3 \times \text{ULN}$ ).

#### **5.1.1.4.3.1 Potential Hy's Law**

Potential Hy's Law criteria will be summarized by treatment group for the Safety Population as follows:

Table 5-22 Potential Hy's Law Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Potential Hy's Law | Number and percentage of participants | Randomization to | Categorical |
| within 24-hour window | with postbaseline assessment of the | End of Study <sup>1</sup> | descriptives |
| | following laboratory parameters based on | | |
| | blood draws collected within a 24-hour | | |
| | period: | | |
| | • ALT or AST $\geq 3 \times ULN$ | | |
| | • TBL $\geq$ 2 × ULN | | |
| | • $ALP < 2 \times ULN$ | | |
| Potential Hy's Law | Number and percentage of participants | Randomization to | Categorical |
| without window | with postbaseline assessment of the | End of Study <sup>1</sup> | descriptives |
| (e-DISH) | following laboratory parameters at any | | |
| | time: | | |
| | <ul> <li>Maximum ALT or AST ≥ 3 ×</li> </ul> | | |
| | ULN | | |
| | • Maximum TBL ≥ 2 × ULN | | |

e-DISH = evaluation of drug-induced serious hepatotoxicity.

Participants who meet the Potential Hy's Law criteria will have their ALT, AST, TBL, and ALP assessment listed for all study visits.

## **5.1.1.4.4 Vital Signs**

Vital signs will be summarized by treatment group for the Safety Population as follows:

Table 5-23 Vital Signs Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| PCS values <sup>1</sup> | Summary of number and percentage of | Randomization to | PCS descriptives |
| | participants by parameter and PCS criteria | End of Study <sup>1</sup> | |
| | <ul> <li>Parameters and PCS criteria specified in</li> </ul> | | |
| | Section 6.3.6.1 | | |
| Descriptives <sup>3</sup> | Summary by parameter and analysis visit | Randomization to | CFB descriptives |
| | <ul> <li>Parameters specified in Section 6.3.6.2</li> </ul> | End of Study <sup>2</sup> | |
| Measures | Summary of number number and percentage of | Randomization to | Summary |

<sup>&</sup>lt;sup>5</sup> Participants with at least one adjudicated case (i.e.  $ALT \ge 3xULN$  or  $AST \ge 3xULN$ ) will be listed with their ALT and AST assessments, adjudication dates, adjudication results and confounding factors for all study visits.

ALT = alanine aminotransferase; AST = aspartate aminotransferase; TBL = total bilirubin.

ALP = alkaline phosphatase; ULN = upper limit of normal.

<sup>&</sup>lt;sup>1</sup> Analysis visits defined in Section 6.2.2.

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| meeting criteria <sup>4</sup> | participants with post-treatment vital sign | End of Study <sup>2</sup> | |
| | measurement meeting any of following criteria | | |
| | will by treatment group: | | |
| | <ul> <li>Systolic Blood Pressure: &lt; 90 mmHg, &gt;</li> </ul> | | |
| | 140 mmHg, > 160 mmHg | | |
| | <ul> <li>Diastolic Blood Pressure: &lt; 50 mmHg, &gt;</li> </ul> | | |
| | 90 mmHg, > 100 mmHg | | |
| | • Pulse Rate: < 60 bpm, > 100 bpm | | |
| | • Temperature: > 38.0 °C, < 36.0 °C | | |
| | • Respiratory rate: < 12 breaths/min, > 20 | | |
| | breaths/min | | |

<sup>&</sup>lt;sup>1</sup> Participants who report ≥ 1 postbaseline PCS value will have their vital sign visits with PCS values and all AEs listed. 
<sup>2</sup> Analysis visits defined in Section 6.2.2.

#### **Electrocardiograms** 5.1.1.4.5

Electrocardiograms (ECGs) will be summarized by treatment group for the Safety Population as follows:

**Table 5-24 ECG Summaries** 

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| PCS values <sup>1</sup> | Summary of number and percentage of participants by parameter and PCS criteria • Parameters and PCS criteria specified in Section 6.3.7.2 • N1 (percentage denominator) = Participants with non-missing non-PCS baseline and >=1 postbaseline parameter assessment | Randomization to<br>End of Study <sup>2</sup> | PCS descriptives |
| Descriptives | <ul> <li>Summary by parameter and analysis visit</li> <li>Parameters specified in Section</li> <li>6.3.7.3</li> </ul> | Randomization to<br>End of Study <sup>2</sup> | CFB descriptives |
| Shift from baseline | <ul> <li>Summary by parameter and category</li> <li>Normal; abnormal, not clinically significant; abnormal, clinically significant provided by investigator</li> <li>Parameters specified in Section 6.3.7.3</li> </ul> | End of Study <sup>2</sup> | Shift analysis |
| Clinically significant<br>ECG abnormalities | A listing showing ECG parameters for participants with postbaseline clinically significant ECG abnormalities according to the investigator's overall interpretation | Randomization to<br>End of Study <sup>2</sup> | Listing |
| Descriptives of measures meeting criteria | Summary of number and percentage of participants with post-treatment QTcF >450 ms, >480 ms, and >500 ms will be tabulated by treatment group | Randomization to<br>End of Study <sup>2</sup> | Descriptives |

Participants who report  $\geq 1$  postbaseline PCS value will have their ECG visits with PCS values and all AEs listed.

<sup>&</sup>lt;sup>3</sup> Participant vital signs will be listed.

<sup>&</sup>lt;sup>4</sup> A listing of AEs for participants with postbaseline values meeting the criteria will be also provided.

<sup>&</sup>lt;sup>2</sup> Analysis visits defined in Section 6.2.2.

#### 5.1.1.4.6 Cardiovascular Risk

Patients will be categorized into 1 of 3 coronary heart disease (CHD) risk subgroups (low, moderate, or high risk) based on NCEP ATP III guideline. Subgroup analyses of TEAEs by cardiovascular (CV) risk category will be provided for the Safety Population.

Table 5-25 Cardiovascular Risk Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| TEAEs | <ul> <li>Subgroup analyses by CV risk</li> </ul> | From randomization | Categorical |
| | category for overall summary and | date to Visit 16 for | descriptives |
| | by SOC and PT | participants with | |
| | | Visit 16, or within | |
| | | 30 days after last | |
| | | visit or last | |
| | | treatment, | |
| | | whichever is later, | |
| | | for participants | |
| | | without Visit 16 | |

#### 5.1.1.4.7 Suicidality Analyses

Suicidality will be summarized by treatment group for the Safety Population as follows:

Table 5-26 Suicidality Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| participants w | number and percentage of ith suicidal ideation and vior for each study phase ming column | Lifetime History, 6<br>months prior to<br>Screening in the<br>lead-in study,<br>Treatment phase,<br>Safety Follow-up<br>phase | Categorical descriptives |

<sup>&</sup>lt;sup>1</sup> Participants with all values, including participant number, treatment group, visit number, intensity of suicidal ideation, suicidal behavior type, and lethality of suicidal behavior will be listed.

#### 5.1.1.5 Subgroup Analyses

Subgroups analyses will be done for disposition (Table 5-6), treatment exposure (Table 5-16), and TEAEs (Table 5-19) for sex, age group ( $<40 \text{ vs} \ge 40$ , and  $<65 \text{ vs} \ge 65$ ), race (White vs. all other races), cardiovascular risk category, and renal function class.

#### 5.1.1.6 Interim Analyses

The interim analysis will occur when at least 300 ubrogepant participants (with a minimum of 2 migraines treated with ubrogepant per month, on average) have been enrolled in the study for 6 months, and 200 ubrogepant participants (with a minimum of 2 migraines treated with ubrogepant per month, on average) have been enrolled in the study for 1 year.

The treatment assignments will be unblinded to the Allergan staff for the interim analyses. The interim analyses will include all analyses specified in this SAP except for efficacy analyses.



# **5.2** Changes in the Conduct of the Study or Planned Analyses

Prior to database lock, there were no changes in study conduct or planned analyses from what was described in the protocol and detailed in the SAP.

#### 5.2.1 Changes in the Conduct of the Study

Not applicable.

### **5.2.2** Changes to Analyses Prior to Database Lock

During study UBR-MD-04, it was reported that Participant attempted to conceal her pregnancy . Therefore, the participant will be excluded from the mITT and safety populations, but will remain in the ITT population. This change is made after interim lock and prior to the final database lock.
# 6. Data Handling and Analysis Conventions

# **6.1 Study Treatment Conventions**

#### 6.1.1 Analysis Days

Treatment day is defined as follows:

Table 6-1 Analysis Day Definitions

| Term | Description |
|---|---|
| Treatment Day | Relative to randomization date |
| | If analysis date ≥ randomization date: |
| | <ul> <li>Day = analysis date - randomization date + 1</li> </ul> |
| | <ul> <li>Day 1 = randomization date</li> </ul> |
| | If analysis date < randomization date: |
| | <ul> <li>Day = analysis date – randomization date</li> </ul> |
| | <ul> <li>Day -1 = day before randomization date</li> </ul> |
| | o There is no Day 0 |

## **6.1.2** Missing/Incomplete Treatment End Date

If the investigator is unable to provide the treatment end date, treatment end date will be imputed to the last available dosing record date.

## 6.2 Analysis Visit Windows



<sup>1</sup>X is 1, 2, 3, ....



# 6.2.2 Safety

The safety analysis visit windows for 3-month time interval are defined as follows:

Table 6-4 Safety Analysis Visit Definitions for 3-Month Time Interval

| <b>Analysis Phase</b> | Analysis Visit (Derived) | Window |
|---|---|---|
| Treatment | Completed 3 months | Treatment Day >= 90 |
| | Completed 6 months | Treatment Day >= 180 |
| | Completed 9 months | Treatment Day >= 270 |
| | Completed 12 months | Completing treatment period per |
| | | disposition CRF, or discontinued |
| | | after day 360 |

Table 6-5 Safety Analysis Visit Definitions for 1-Month Time Interval

| Analysis Phase | Analysis Visit (Derived) | Window |
|----------------|--------------------------------|----------------------------|
| Treatment | Months 1 Treatment Day [1, 30] | |
| | Months 2 | Treatment Day [31, 60] |
| | Months 3 | Treatment Day [61, 90] |
| | Months 4 | Treatment Day [91, 120] |
| | Months 5 | Treatment Day [121, 150] |
| | Months 6 | Treatment Day [151, 180] |
| | Months 7 | Treatment Day [181, 210] |
| | Months 8 | Treatment Day [211, 240] |
| | Months 9 | Treatment Day [241, 270] |
| | Months 10 | Treatment Day [271, 300] |
| | Months 11 | Treatment Day [301, 330] |
| | Months 12 | Treatment Day [331, end of |
| | | treatment period] |

The analysis visit windows for safety endpoints are defined as follows:

Table 6-6 Safety Analysis Visit Definitions

| <b>Analysis Phase</b> | Analysis Visit (Derived) | Scheduled Study Visit (eCRF) | Window |
|---|---|---|---|
| Pretreatment | Baseline | Baseline from Lead-in Study | Treatment Day ≤ 1 |
| | Week 4 | (Visit 3) Week 4 | Treatment Day [2, 42] |
| | Week 8 | (Visit 4) Week 8 | Treatment Day [43, 70] |
| | Week 12 | (Visit 5) Week 12 | Treatment Day [71, 98] |
| | Week 16 | (Visit 6) Week 16 | Treatment Day [99, 126] |
| | Week 20 | (Visit 7) Week 20 | Treatment Day [127, 154] |
| | Week 24 | (Visit 8) Week 24 | Treatment Day [155, 182] |
| | Week 28 | (Visit 9) Week 28 | Treatment Day [183, 210] |
| | Week 32 | (Visit 10) Week 32 | Treatment Day [211, 238] |
| | Week 36 | (Visit 11) Week 36 | Treatment Day [239, 266] |
| | Week 40 | (Visit 12) Week 40 | Treatment Day [267, 294] |
| | Week 44 | (Visit 13) Week 44 | Treatment Day [295, 322] |
| | Week 48 | (Visit 14) Week 48 | Treatment Day [323, 350] |
| | Week 52 | (Visit 15) Week 52/Early | Treatment Day [351, end of |
| | | Termination | treatment period] |

| <b>Analysis Phase</b> | Analysis Visit (Derived) | Scheduled Study Visit (eCRF) | Window |
|---|---|---|---|
| | Safety Follow-up | (Visit 16) 4 Week Safety | Treatment Day [end of treatment |
| | | Follow-up | period+1, the last study visit] |
| | End of study | Final or termination visit | Latest non-missing assessment |
| | - | | after randomization date |

Safety follow-up visit will be presented in analysis tables for clinical laboratory values and vital signs. End of Study is defined as the last available assessment during treatment and/or safety follow-up period. End of Study results will be presented in analysis tables for safety parameters, including but not limited to electrocardiograms, clinical laboratory values, and vital signs.

The following general conventions for repeated or unscheduled assessments will apply unless otherwise specified:

- The latest non-missing assessment within any analysis window will be flagged as the analysis value for any summaries by analysis visit
- All postbaseline assessments will be considered for PCS categorization
- All assessments will be included in respective listings







# **6.3.4.2 AE** Group of Interest

The preferred terms included in each category are based on standardized MedDRA queries (SMQs) or are custom created where no SMQ exists or is inadequate (as shown in Table 6-10).

**Table 6-10** Construction Methods for AE Categories of Clinical Interest

| Method | Category |
|---|---|
| | Cardiac arrhythmias |
| | Arrhythmia related investigations, signs and symptoms |
| | • Cardiac arrhythmia terms (incl bradyarrhythmias and tachyarrhythmias) Central nervous system vascular disorders |
| | <ul> <li>Central nervous system haemorrhages and cerebrovascular conditions</li> <li>Central nervous system vascular disorders, not specified as haemorrhagic or ischaemic</li> </ul> |
| | Embolic and thrombotic events |
| Narrow SMQs | Embolic and thrombotic events, arterial |
| | <ul> <li>Embolic and thrombotic events, venous</li> <li>Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous</li> <li>Hypertension</li> </ul> |
| | Ischaemic heart disease |
| | Myocardial infarction |
| | Other ischaemic heart disease Suicide/self-injury |
| | Hepatic injury |
| | Hepatic disorders (broad SMQ) |
| Custom created | • Liver transplant (preferred term) Abuse-related |
| | Triptan-associated |

| Method | Category |
|--------|----------|

Note: the categories of clinical interest are listed in bolded italics fonts and constructed from Standard MedDRA Query Version 20.1.

The preferred term for the custom-created abuse-related category and triptan-associated category are provided in Table 6-11. The lists of preferred terms for AE categories of clinical interest created using SMQs are provided in Appendix I.

Table 6-11 Preferred Terms for Abuse-Related Category and Triptan-Associated Category

| Category | Preferred Terms |
|---|---|
| Triptan Associated | chest pain; chest discomfort; throat tightness; asthenia; paraesthesia; dysaesthesia; hyperaesthesia |
| Abuse Related | Affective disorder; Aggression; Confusional state; Disorientation; Dizziness; Drug tolerance; Drug withdrawal syndrome; Euphoric mood; Feeling abnormal; Feeling drunk; Feeling of relaxation; Hallucination; Inappropriate affect; Mood altered; Psychotic disorder; Somnolence; Substance abuse; Substance dependence; Substance use; Substance-induced mood disorder; Substance-induced psychotic disorder; Thinking abnormal |

#### 6.3.5 Clinical Laboratory Assessments

# **6.3.5.1** Potentially Clinically Significant Criteria

Laboratory assessments values meeting *any* of the following PCS low or PCS high criteria will be categorized as PCS:

Table 6-12 Clinical Laboratory PCS Criteria

| Laboratory<br>Group | Parameter | SI Unit | PCS Low<br>Limit | PCS High<br>Limit |
|---|---|---|---|---|
| _ | Basophils, absolute cell count | 10 <sup>9</sup> /L | _ | > 2.0 × ULN |
| | Eosinophils absolute cell count | 10 <sup>9</sup> /L | _ | > 2 × ULN |
| | Hematocrit | Ratio | < 0.9 × LLN | > 1.1 × ULN |
| | Hemoglobin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Lymphocytes absolute cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.3 × ULN |
| Hematology | Monocytes, absolute cell count | 10 <sup>9</sup> /L | < 0.5 × LLN | > 2.0 × ULN |
| | Neutrophils absolute cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.3 × ULN |
| | Platelet count (thrombocytes) | 10 <sup>9</sup> /L | < 0.5 × LLN | > 1.5 × ULN |
| | Red blood cell count | 10 <sup>12</sup> /L | < 0.9 × LLN | > 1.1 × ULN |
| | White blood cell count | 10 <sup>9</sup> /L | < 0.9 × LLN | > 1.5 × ULN |
| Chemistry | Alanine aminotransferase | U/L | _ | > 3 × ULN |
| Chemistry | Albumin | g/L | < 0.8 × LLN | > 1.2 × ULN |

| Laboratory<br>Group | Parameter | | PCS Low<br>Limit | PCS High<br>Limit |
|---|---|---|---|---|
| | Alkaline phosphatase | U/L | _ | > 3 × ULN |
| | Aspartate aminotransferase | U/L | _ | > 3 × ULN |
| | Bicarbonate | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Bilirubin, total | μmol/L | _ | > 1.5 × ULN |
| | Blood urea nitrogen | mmol/L | _ | > 1.5 × ULN |
| | Calcium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Chloride | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Cholesterol, total | mmol/L | _ | > 1.6 × ULN |
| | Creatinine | μmol/L | _ | > 1.5 × ULN |
| | Creatine kinase | | _ | > 2.0 × ULN |
| | Glucose, nonfasting | mmol/L | < 0.8 × LLN | > 2 × ULN |
| | Lactate dehydrogenase (LDH) | U/L | _ | > 3.0 × ULN |
| | Phosphorus | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Potassium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Protein, total | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Sodium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Triglycerides | mmol/L | _ | > 2.0 × ULN |
| | Uric acid (urate) | μmol/L | _ | > 1.2 × ULN |
| | Glucose | mmol/L | | Positive |
| Urinolygia | рН | рН | < 0.9 × LLN | > 1.1 × ULN |
| Urinalysis | Protein | g/L | _ | Positive |
| | Specific gravity | | | > 1.1 × ULN |

LLN = lower limit of normal (value provided by the laboratory); PCS = potentially clinically significant; SI = *Le Système International d'Unités* (International System of Units); ULN = upper limit of normal (value provided by the laboratory).

# **6.3.5.2** Hepatic Laboratory Abnormalities

The selected event is of clinical interest: Elevated ALT or AST lab value that is  $\geq 3$  times the ULN. The following laboratory parameters will be summarized:

Table 6-13 Criteria for Hepatic Laboratory Abnormalities

| Laboratory Parameter | Categories |
|----------------------|--------------|
| | >= 1 × ULN |
| | >= 1.5 × ULN |
| | >= 2 × ULN |
| ALT | >= 3 × ULN |
| | >= 5 × ULN |
| | >= 10 × ULN |
| | >= 20 × ULN |
| | >= 1 × ULN |
| | >= 1.5 × ULN |
| | >= 2 × ULN |
| AST | >= 3 × ULN |
| | >= 5 × ULN |
| | >= 10 × ULN |
| | >= 20 × ULN |
| ALT or AST | >= 1 × ULN |
| | >= 1.5 × ULN |
| | >= 2 × ULN |
| | >= 3 × ULN |
| | >= 5 × ULN |
| | >= 10 × ULN |
| | >= 20 × ULN |
| | >= 1 × ULN |
| | >= 1.5 × ULN |
| | >= 2 × ULN |
| Bilirubin Total | >= 3 × ULN |
| | >= 5 × ULN |
| | >= 10 × ULN |
| | >= 20 × ULN |
| | >= 1 × ULN |
| | >= 1.5 × ULN |
| Alkaline Phosphatase | >= 2 × ULN |
| | >= 3 × ULN |
| | >= 5 × ULN |

| Laboratory Parameter | Categories |
|---|---|
| | >= 10 × ULN |
| | >= 20 × ULN |
| Concurrent Elevations <sup>1</sup> | ALT or AST $\geq$ = 3 × ULN <b>AND</b> Bilirubin Total $\geq$ 1.5 × ULN |
| Concurrent Elevations | ALT or AST $>= 3 \times ULN$ <b>AND</b> Bilirubin Total $\geq 2 \times ULN$ |
| Potential Hy's Law <sup>1</sup> | ALT or AST $\geq$ 3 × ULN <b>AND</b> Bilirubin Total $\geq$ 2 × ULN AND ALP < 2 × ULN |

LLN = lower limit of normal (value provided by the laboratory); PCS = potentially clinically significant; SI = Le Système International d'Unités (International System of Units); ULN = upper limit of normal (value provided by the laboratory).

#### 6.3.5.3 Continuous Descriptives and Shift Table Parameters

The following laboratory parameters will be summarized:

Table 6-14 Clinical Descriptive and Shift Table Parameters

| Category | Parameters |
|---|---|
| Chemistry | Sodium, potassium, chloride, bicarbonate, glucose, blood urea nitrogen, creatinine, total |
| | bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, |
| | lactate dehydrogenase, creatine kinase, total protein, albumin, calcium, phosphorus, uric |
| | acid, total cholesterol, high density lipoprotein, low density lipoprotein, total |
| | triglycerides |
| Hematology | Hemoglobin; hematocrit; red blood cell count; red blood cell indices (mean corpuscular |
| | volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration); |
| | white blood cell count, including differential (neutrophils, lymphocytes, monocytes, |
| | eosinophils, and basophils); platelet count |
| Urinalysis | Specific gravity, pH |

#### 6.3.5.4 Character Values

Character values (eg, < 5, negative) will be reviewed prior to database lock and converted to numeric for analysis as appropriate. These conversions will be documented in the ADaM specifications.

#### 6.3.6 Vital Signs

# 6.3.6.1 Potentially Clinically Significant Criteria

Vital sign values meeting *both* the actual value and change from baseline PCS criteria will be categorized as PCS:

Table 6-15 Vital Sign PCS Criteria

| Vital Sign | Flag | Criterion Value | Change From Baseline or<br>Predose |
|---|---|---|---|
| Systolic blood pressure, mm Hg | High | ≥ 180 | Increase of ≥ 20 |
| Systolic blood pressure, fillit rig | Low | ≤ 90 | Decrease of ≥ 20 |
| Diastolic blood pressure, mm Hg | High | ≥ 105 | Increase of ≥ 15 |

<sup>&</sup>lt;sup>1</sup> Elevations are from the same day

| | Low | ≤ 50 | Decrease of $\geq 15$ |
|------------------------------------|------|-------|------------------------|
| Pulsa rata ham | High | ≥ 120 | Increase of $\geq 15$ |
| Pulse rate, bpm | Low | ≤ 50 | Decrease of $\geq 15$ |
| Weight, kg | High | _ | Increase of $\geq 7\%$ |
| weight, kg | Low | | Decrease of ≥ 7% |
| Orthostatic SBP change, mm Hg | Low | ≤ -20 | |
| Orthostatic DBP change, mm Hg | Low | ≤-15 | |
| Orthostatic Pulse rate change, bpm | High | ≥ 25 | |

SBP = Systolic blood pressure, DBP = Diastolic blood pressure, bpm = beats per minute.

## 6.3.6.2 Continuous Descriptives and Shift Table Parameters

The following vital sign parameters will be summarized:

Table 6-16 Vital Sign Descriptive and Shift Table Parameters

| Parameters | | |
|---|---|---|
| SBP | Respiratory rate | Weight |
| DBP | Temperature | BMI |
| Pulse rate | Orthostatic SBP changes <sup>1</sup> | Orthostatic DBP change <sup>1</sup> |
| Orthostatic Pulse rate change <sup>1</sup> | | |

SBP = Systolic blood pressure. DBP = Diastolic blood pressure. BMI=Body Mass Index.

## 6.3.7 Electrocardiograms

#### **6.3.7.1 QTc Derivation**

QTc Bazett (QTcB) and QTc Fridericia (QTcF) are derived as follows:

**Table 6-17 QTc Derivation** 

| Parameter | Derivation if RR available | Derivation if RR unavailable |
|-----------|----------------------------|------------------------------|
| QTcB | QT | QT |
| | square root of RR | square root of (60/HR) |
| QTcF | QT | QT |
| | cubic root of RR | cubic root of (60/HR) |

QTcB = QTc Bazett; QTcF = QTcF Fridericia.

## 6.3.7.2 Potentially Clinically Significant Criteria

ECG values meeting *either* the actual value or change from baseline PCS high criteria will be categorized as PCS:

<sup>&</sup>lt;sup>1</sup>Orthostatic pulse rate change equals standing pulse rate minus sitting pulse rate; orthostatic systolic blood pressure change equals standing systolic blood pressure minus sitting systolic blood pressure; and orthostatic diastolic blood pressure change equals standing diastolic blood pressure minus sitting diastolic blood pressure

Table 6-18 ECG PCS Criteria

| Parameter | Unit | Criterion Value | Change from Baseline or<br>Predose |
|---|---|---|---|
| QRS duration | msec | ≥ 150 | _ |
| PR interval | msec | ≥ 250 | _ |
| QTc (QTcB or QTcF) interval | msec | > 500 | Increase of > 60 |

PCS = potentially clinically significant; QTc = corrected QT interval QTcB = QTc Bazett; QTcF = QTcF Fridericia.

#### 6.3.7.3 Continuous Descriptives and Shift Table Parameters

The following ECG parameters will be summarized:

Table 6-19 ECG Descriptive and Shift Table Parameters

| Parameters | | |
|-------------------------------------|------------------|------|
| Heart rate QRS interval QT interval | | |
| | PR interval | QTcB |
| | RR interval QTcF | |

QTcB = QTc Bazett; QTcF = QTcF Fridericia.

#### 6.4 Imputed Value Listing Conventions

In general, listings will present the actual partial or missing values rather than the imputed values that may be used in endpoint derivation. In instances where imputed values will be presented, imputed values will be flagged. Actual rules will be fully defined in the table, figure, and data listing specification document

# 7. Amendment(s)

In Section 5.1.1.4.2, removed triptan-associated and abuse-related AE from Table 5-19, for Table 5-20, triptan-associated and abuse-related TEAE were under TEAE of special interest.

In Table 5-20 (Section 5.1.1.4.2), removed Triptan-associated TEAE from the overall summary row.

In Table 6-4 (Section 6.2.2), updated definition of completing 12 months.

Added details of AE group of special interest (Section 6.3.4.2).

Added Appendix I: Preferred Terms for AE Categories of Clinical Interest Created by SMQs (Section 8.1).

In Section 5.1.1.4.2 added additional analyses of TEAE reported in  $\geq$  2% of participants in any ubrogepant treated dose group (and greater than placebo) sorted by SOC and then by Preferred Term.

In Section 5.1.1.4.4 added additional analyses of vital signs for measures meeting criteria.

In Section 5.1.1.4.5 added additional analyses of ECG for measures meeting criteria.

In Section 6.4.4, imputation method is changed, missing AE will not be imputed. Updated the imputation of medication end date in case imputed end date is prior to start date, the end date will be imputed the same as the start date.

# 8. Appendices

# 8.1 Appendix I: Preferred Terms for AE Categories of Clinical Interest Created by SMQs.

Table 8-1 List of Preferred Terms for AE Categories of Clinical Interest Created by Narrow SMQs.


| Category | Subcategory | SMQ Type | Preferred Term |
|----------|-------------|----------|--------------------------|
| | | Narrow | Subendocardial ischaemia |

Table 8-2 List of Preferred Terms for Hepatic Disorder Broad SMQ

